CLINICAL TRIAL: NCT03574688
Title: The Hydration to Optimize Metabolism (H2O Metabolism) Pilot Study
Acronym: H2OMetaboPilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Olle Melander, Professor, Region Skane
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016894_PILOT
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Low Water Intake; High Vasopressin
Keywords: Hydration; Water; Vasopressin; Copeptin; Glucose
MeSH Terms: conditions — Diabetes Insipidus | interventions — Water

STUDY DESIGN:
Intervention Model Description: All participants of this pilot intervention study had the intervention of 1.5 Liters of increased daily water intake per day during 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Water intervention (Experimental): The participants increase their habitual daily water intake with 1.5 Liters of tap water per day during 6 weeks.
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Water — Increased daily water intake with 1.5 Liters of water per day on top of habitual water intake.

SUMMARY:
This study evaluates increased hydration (1.5 L of water daily during 6 weeks) on top of habitual water intake in the lowering of the vasopressin marker copeptin and in the lowering of plasma glucose concentration in adults with signs of low water intake at recruitment (elevated levels of copeptin, high urine osmolality, low urine volume).

DETAILED DESCRIPTION:
High plasma concentration of vasopressin (i.e. antidiuretic hormone) is a novel and independent risk factor for type 2 diabetes, the metabolic syndrome, cardiovascular disease and premature death. The main physiological role of vasopressin is to maintain constant plasma osmolality. Previous studies in rats and a Mendelian randomization study in humans suggest causality between elevated vasopressin concentration and elevated plasma glucose concentration. As vasopressin can be suppressed by increasing water intake, the investigators hypothesize that water supplementation in individuals with high vasopressin can lower plasma glucose and prevent diabetes.

The aim of this pilot study is to test if six weeks of water supplementation of 1.5 Liters of extra water per day in low-drinkers with high copeptin can significantly alter hydration markers in general and reduce plasma copeptin in particular. Furthermore, the investigators also aim at investigating whether this 6-week water intervention can significantly reduce fasting plasma glucose concentration.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Age 20-75 years
* High plasma concentration of copeptin of >6.1 pmol/L in women and > 10.7 pmol/L in men
* 24-hour urine osmolality > 600 milliosmol (mosm) /kg water.

Exclusion Criteria:

* 24-hour urine volume >1.5 L
* Pregnancy or breastfeeding
* Plasma sodium <135 mmol/L
* Use of diuretics, lithium or SSRI drugs
* Chronic kidney disease (estimated glomerular filtration rate < 30mL/min)
* Heart failure
* Inflammatory bowel disease
* Type 1 diabetes or type 2 diabetes treated with insulin
* Vulnerable subjects (subjects with legal guardian, with loss of personal liberty)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Fasting plasma copeptin concentration (pmol/L) | 6 weeks
  Change of fasting plasma copeptin between baseline and after 6 weeks of increased water intake.

SECONDARY OUTCOMES:
24 hour urine osmolality (mosm/kg H2O) | 6 weeks
  Change of 24 hour urine osmolality between baseline and after 6 weeks of increased water intake.
24 hour urine volume (L/24h) | 6 weeks
  Change of 24 hour urine volume between baseline and after 6 weeks of increased water intake.
Drinking water (L/day) | 6 weeks
  Change of intake of tap and bottled water between baseline and after 6 weeks of increased water intake.
Total water (L/day) | 6 weeks
  Change of total water intake between baseline and after 6 weeks of increased water intake.
Fasting plasma glucose concentration (mmol/L) | 6 weeks
  Change of Fasting plasma glucose concentration between baseline and after 6 weeks of increased water intake.

CONTACTS AND LOCATIONS:
Overall Officials: Olle Melander, M.D., Prof, Principal Investigator — Lund University
Locations (1):
- KFE, Skåne University Hospital in Malmö, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Enhorning S, Vanhaecke T, Dolci A, Perrier ET, Melander O. Investigation of possible underlying mechanisms behind water-induced glucose reduction in adults with high copeptin. Sci Rep. 2021 Dec 29;11(1):24481. doi: 10.1038/s41598-021-04224-5. PMID 34966186
- [Derived] Enhorning S, Brunkwall L, Tasevska I, Ericson U, Persson Tholin J, Persson M, Lemetais G, Vanhaecke T, Dolci A, Perrier ET, Melander O. Water Supplementation Reduces Copeptin and Plasma Glucose in Adults With High Copeptin: The H2O Metabolism Pilot Study. J Clin Endocrinol Metab. 2019 Jun 1;104(6):1917-1925. doi: 10.1210/jc.2018-02195. PMID 30566641

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT03574688/Prot_SAP_000.pdf